CLINICAL TRIAL: NCT00638118
Title: A Comparison of Fexofenadine HCl 180 mg, Montelukast Sodium 10 mg and Placebo in Suppression of Wheal and Flare Induced by Seasonal Allergen
Brief Title: Fexofenadine HCl 180 mg, Montelukast Sodium 10 mg and Placebo in Suppression of Wheal and Flare Induced by Seasonal Allergen
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Study Director, sanofi-aventis
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: M016455A_4146
Record Dates: First submitted 2008-03-10; First posted 2008-03-18 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2011-01

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — fexofenadine

INTERVENTIONS:
Drug: Fexofenadine

SUMMARY:
Examine the relative potency, onset of action and duration of action of fexofenadine HCl 180 mg (Allegra) and montelukast sodium 10 mg (Singulair) as compared to placebo on skin wheals and flares induced by seasonal allergen.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, 15 to 55 years of age, may participate.
* Subjects with a history of seasonal allergic rhinitis (due to ragweed; oak, elm or maple; or grasses) for the previous 2 years.
* Positive seasonal allergen skin prick tests (or duplicate seasonal allergen skin prick test) with a summation flare greater than or equal to 20 mm larger than diluent control, and summation wheal greater than or equal to 6 mm larger than diluent control at the screening visit 1 (see Appendix 17.1); the seasonal allergen testing that results in the greatest summation flare will be used for all subsequent seasonal allergen testing.
* All female subjects must have a negative urine pregnancy test at the screening visit.
* Female subjects who are sexually active will be expected to use one of the following birth control methods throughout the study.
* Subjects must be within 15% of normal body weight for height or a BMI less than 29.9 (based on NHLBI guidelines).
* Subjects willing and able to adhere to visit schedules and all study requirements.
* All female subjects must have a negative urine pregnancy test at each treatment visit (Visit 2, 4, and 6).
* Continues to meet all inclusion and exclusion criteria.

Exclusion Criteria:

* Asthma that requires treatment with medication other than an inhaled, short-acting beta agonist.
* Significant signs and symptoms of currently active allergic disease (SAR, perennial allergic rhinitis, episodic allergic rhinitis).
* Upper respiratory tract infection, sinusitis, asthma or flu-like symptoms within 2 weeks prior to visit 1.
* Subjects who have dermatographism or other skin conditions which might interfere with the interpretation of the skin test results.
* Subjects who are receiving escalating doses of immunotherapy, oral immunotherapy or short course (rush) immunotherapy.
* Any excessive amounts of alcohol (no more than two drinks/day on average).
* Any excessive use of caffeine (more than six cups of coffee per day or equivalent).
* Any history of chronic alcohol or mood-altering drug abuse.
* Any use of tobacco/nicotine products within 90 days of visit 1.
* Any disease state or surgery known to affect the gastrointestinal absorption of drugs.
* Known hypersensitivity to the investigational product or to drugs with similar chemical properties.
* Subjects who will be visiting a tanning salon during the study.
* Subjects who will need to use artificial tanning products during the study.
* Pregnancy.
* Breast-feeding.
* Regular treatment with other H1-receptor antagonists in the last year before study entry.
* No person or child of a person directly associated with the administration of the study may participate as a study subject.
* Likelihood of requiring treatment during the study period with drugs not permitted by the clinical study protocol.
* Treatment with any investigational product in the last 30 days before study entry.
* Clinically relevant cardiovascular, hepatic, neurologic, endocrine, or other major systemic disease making implementation of the protocol or interpretation of the study results difficult.
* Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study.
* Subject unlikely to comply with protocol, e.g., uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study.
* Use of any of the following drugs within the time indicated prior to the first dosing visit: Systemic or injected corticosteroids (including oral, parenteral, intravenous, rectal) 30 days; Nasal or inhaled or ocular corticosteroids 30 days; Nasal or inhaled ipratropium bromide (or atropine), inhaled nedocromil, or nasal, inhaled, or ophthalmic sodium cromolyn 14 days; Agents with antihistaminic/anticholinergic activity (e.g. antidepressants, antipsychotics) 14 days; Leukotriene pathway modifiers (Accolate, Singulair, Zyflo) 10 days; Ocular anti-allergy medications including lodoxamide (Alomide), olopatadine (Patanol), emedastine difumarate (Emadine), levocabastine (Livostin) 10 days; Non-steroidal anti-inflammatory ophthalmics including ketorolac (Acular), flurbiprofen (Ocufen), suprofen (Profenal), diclofenac (Voltaren) 10 days; Antihistamines including desloratadine (Clarinex), loratadine (Claritin) 10 days; Antihistamines including fexofenadine HCl (Allegra), cetirizine (Zyrtec), hydroxyzine, azelastine nasal spray (Astelin), clemastine 7 days; Other short-acting antihistamines such as chlorpheniramine or drugs with antihistaminic activity 3 days; OTC oral antihistamines, decongestants (includes pseudoephedrine and other decongestants), or antihistamines/decongestant combinations including all cold, cough, and sleep aids 3 days; OTC ophthalmic decongestant,antihistamine, or decongestant/antihistamine combinations 3 days; Other anticholinergic agents 3 days; Immunotherapy injection 1 day.
* Other drugs should only be permitted if they are not expected to interfere with the ability of the subject to participate in the study.
* Non-steroidal anti-inflammatory agents are not allowed for 2 days prior to each treatment visit day through 25 hours post-dose (low-dose cardiac prophylaxis is allowed).
* Use of any medications or agents that are not specified above that may confound the interpretation of the results:
* Caffeine within 6 hours prior to each visit (coffee, tea, cola, and sodas, including Mountain Dew and Surge)
* Decaffeinated coffee, tea and colas within 6 hours of each visit
* Alcohol within 24 hours prior to each study visit
* Chocolate within 6 hours prior to each visit
* Antacids within +/- minus2 hours of investigational product dosing.

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2003-02; Study Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
Size of change in skin flares from baseline will be measured. | Post-dose (20 min, 40 min, 60 min, and hourly through 12 hours with an additional 2 time points obtained at Hours 23 and 24)

SECONDARY OUTCOMES:
Size of change in skin wheals from baseline will be measured. | Post-dose (20 min, 40 min, 60 min, and hourly through 12 hours with an additional 2 time points obtained at Hours 23 and 24)

CONTACTS AND LOCATIONS:
Overall Officials: Phyllis Diener, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Bridgewater, New Jersey, United States